CLINICAL TRIAL: NCT00233493
Title: Demonstration of the Spread of Dermatophytes Through Casual Contact Among Family Household Members
Brief Title: Spread of Dermatophytes Among Families
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: CSFO327KUS16
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Results first posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-08

CONDITIONS: Onychomycosis; Tinea Pedis
Keywords: dermatophytes
MeSH Terms: conditions — Onychomycosis; Tinea Pedis

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective is to demonstrate person-to-person spread of dermatophytes of the skin and nails among family members, as measured by fungal culture and DNA typing of the dermatophytes isolated.

DETAILED DESCRIPTION:
Enrolled families consist of at least two members over the age of 14. Once the index person is examined and a dermatophyte is isolated from either toenail or foot scale, other family members are examined and cultured. All dermatophyte isolates obtained from each family unit are compared using DNA typing and restriction length polymorphism (RFLP) to determine whether family members share the same organism or were infected by an outside source.

ELIGIBILITY:
Inclusion Criteria: positive dermatophyte culture

-

Exclusion Criteria:

* use of antifungal agents, either oral or topical

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study Design-Households with at least 2 residents and 1 individual (index person [IP]) with tinea pedis and/or onychomycosis were identified by screening. Infection was confirmed clinically and mycologically (potassium hydroxide [KOH] and culture positive) in the IP; then other members within the same household were examined for tinea pedis and/or onychomycosis using the same criteria. All participants with confirmed fungal infections were referred to their primary care physicians for appropriate treatment.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2005-03; Primary Completion 2009-01 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud A Ghannoum, PhD, Principal Investigator — Center for Medical Mycology, University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Households
Groups:
- One Infected Member: One infected member in multiple person household
- 2 or More Infected Members: Two or more infected members in a multiple person household
Period: Overall Study
Arm/Group | One Infected Member | 2 or More Infected Members
Started | 32; 32 Households | 18; 18 Households
Completed | 32; 32 Households | 18; 18 Households
Not Completed | 0; 0 Households | 0; 0 Households

BASELINE CHARACTERISTICS:
Groups:
- Single Person Households: Households with at least 1 resident with tinea pedis and/or onychommycosis.
- Multiperson Households: Households with at least 2 residents and 1 individual with tinea pedis and /or onychommycosis.
- Total: Total of all reporting groups
Arm/Group | Single Person Households | Multiperson Households | Total
Number analyzed (Participants) | 32 | 18 | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.73 (17.61) | 50.33 (20.80) | 54.03 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 6 | 33
  Male | 5 | 12 | 17
Region of Enrollment [Number; unit: participants]
  United States | 32 | 18 | 50

OUTCOME MEASURES:

1. Primary Outcome: Dermatophyte Species Distribution
Description: To identify dermatophytes isolates known to cause onychomycosis and/or tinea pedis by Polymerase Chain Reaction (PCR)
Time Frame: Baseline
Measure: Number; unit: isolates
Units Other Than Participants: Households
Groups:
- SIM Households: SIM Households in which dermatophyte isolates were isolated
- MIM Households: MIM Households in which dermatophyte isolates were identified
Arm/Group | SIM Households | MIM Households
Number analyzed (Participants) | 32 | 18
Number analyzed (Households) | 32 | 18
isolates
  T Rubrum Isolates | 50 | 37
  T Mentagrophytes Isolates | 5 | 12
  E Floccosum Isolates | 2 | 1

2. Secondary Outcome: Dermatophyte Strain Types Among All Enrolled Households
Description: Using southern blot analysis and RFLP to evaluate the isolates and strain types obtained from all enrolled households
Time Frame: Baseline
Measure: Number; unit: isolates
Units Other Than Participants: Households
Groups:
- SIM Households: Isolates obtained from SIM households
- MIM Households: Isolates obtained from MIM households
Arm/Group | SIM Households | MIM Households
Number analyzed (Participants) | 32 | 18
Number analyzed (Households) | 32 | 18
isolates
  T rubrum strain type | 50 | 37
  T mentagrophytes strain types | 5 | 12
  E Floccosum strain types | 2 | 1

3. Secondary Outcome: Number of Households With Dermatophyte Infection Spread
Description: To determine if dermatophyte infection in household members could spread to other members, we analyzed the Southern blot and RFLP band patterns for different clinical isolates obtained from members residing in the same MIM households.
Time Frame: Baseline
Population: This outcome measure was intended to identify the number of households with dermatophyte infection spread in multiple infected member households only.
Measure: Number; unit: Households
Units Other Than Participants: Households
Groups:
- MIM Household: Number of households associated with spread of infection associated with specific strain types
Arm/Group | MIM Household
Number analyzed (Participants) | 18
Number analyzed (Households) | 18
Households
  Spread of Infection due to T Rubrum Isolates | 7
  Spread of Infection due to T Mentagrophytes Isolates | 1
  No Spread of Infection | 10

4. Secondary Outcome: Number of Participants Affected by the Association of Spread of Infection and History of Tinea Pedis or Onychomycosis
Description: The relationship between spread of infection and whether a subject previously had onychomycosis, tinea pedis, or onychomycosis plus tinea pedis was investigated. We collected how many subjects had spread of infection and onychomycosis alone, or spread of infection and tinea pedis alone, as well as how many subjects had spread of infection and onychomycosis plus tinea pedis.
Time Frame: Baseline
Measure: Number; unit: participants
Units Other Than Participants: Households
Groups:
- MIM Household; SIM Household: Host associated factors and spread of infection among individuals residing in the same household
Arm/Group | MIM Household | SIM Household
Number analyzed (Participants) | 32 | 18
Number analyzed (Households) | 32 | 18
participants
  Spread of Infection and history of tinea pedis or onychomycosis | 0 | 0
  Spread of Infection and history of both tinea pedis and onychomycosis | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Event data was not collection, this was a single clinic visit.
Description: Averse Event data was not collected.
Groups:
- Multi Person Households: Households with at least 2 residents and 1 individual with tinea pedis and/or onychomycosis
- Single Person Household: Households with 1 resident/individual with tinea pedis and/or onychomycosis
Arm/Group | Multi Person Households | Single Person Household
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
A cross-sectional, not longitudinal, analysis; therefore, we were unable to determine the chronology of infection, the cause-and-effect relationship between specific strain types and infection, or the household member that was infected first.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No